CLINICAL TRIAL: NCT00909558
Title: A Phase I Open Label, Single Site, Safety and Efficacy Study of the Effects of Autologous Natural Killer and Natural Killer T Cell Immunotherapy on Malignant Disease
Brief Title: Safety and Effectiveness Study of Autologous Natural Killer and Natural Killer T Cells on Cancer
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: Envita Medical Center, Inc. (Industry)
Responsible Party: Santo Prato, N.M. / President, Envita Medical Center, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E001-08
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer; Glioma; Hepatocellular Cancer; Squamous Cell Lung Cancer; Pancreatic Cancer; Colon Cancer; Prostate Cancer
Keywords: metastatic malignancies; tumor markers; chemotherapy; cancer; breast cancer; glioma; hepatocellular cancer; squamous cell lung cancer; pancreatic cancer; colon cancer; prostate cancer
MeSH Terms: conditions — Breast Neoplasms; Glioma; Liver Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Autologous Natural Killer / Natural Killer T Cell Immunotherapy — The study drug is derived from ex vivo expansion of each subject's own white blood cells and is therefore autologous.
  The current study proposes a 3-course treatment of doses administered at one week intervals with monitoring at each administration plus 2 weeks after the last dose. The total study time (apheresis through last follow-up) is estimated at 15 weeks.

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of natural killer (NK) cell and natural killer T (NKT) cell-based autologous adoptive immunotherapy in subjects with metastatic, treatment-refractory breast cancer, glioma, hepatocellular carcinoma, squamous cell lung cancer, pancreatic cancer, colon cancer or prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female not less than 18 years of age or over 80 years of age.
* Life expectancy of ≥ 24 weeks as measured by the Eastern Cooperative Oncology Group (ECOG) performance status.
* Subjects must present with one of the following disease pathologies: Breast Cancer, Glioma, Hepatocellular Cancer, Squamous Cell Lung Cancer, Pancreatic Cancer, Colon Cancer or Prostate Cancer
* The pathology must be an assessable disease (measurable by CT scan or MRI) that is refractory to standard treatments (e.g., chemotherapy, radiation, etc.)
* Negative for hepatitis B, hepatitis C, HIV, and CMV.
* Subjects must present with leukocyte counts above 3,000/μL and platelet counts above 100,000/ μL.
* Subjects must present with minimum hemoglobin levels of 10.
* If female, subject is surgically sterile (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), post menopausal (no menses >12 months), or using a high-efficiency method of contraception such as implant, injectable, combination oral contraceptive, intrauterine device (IUD) or sexual abstinence, or has a vasectomized partner.
* If female of childbearing potential, subject is not pregnant, breast-feeding or planning a pregnancy during the study, and has a negative pregnancy test on screening visit.
* Able to comprehend and sign an informed consent document and comply with the requirements of the study.

Exclusion Criteria:

* No measurable malignant disease by CT scan or tumor markers.
* Life expectancy of ≤ 24 weeks as measured by the Eastern Cooperative Oncology Group (ECOG) performance status.
* Age of less than 18 years or over 80 years of age.
* Documented/confirmed positive testing for hepatitis B, hepatitis C, HIV, or CMV.
* Prior or current history of autoimmune disease.
* Pregnant or lactating women.
* Leukocyte count < 3,000 /μL prior to leukapheresis.
* Platelet count < 100,000/μL prior to leukapheresis.
* Hemoglobin levels below 10.
* PTT (prothrombin time) of < 12 seconds or > than 15 seconds.
* aPTT (activated partial thromboplastin time) of < 25 seconds or > than 39 seconds.
* Failure or refusal to sign informed consent for the study.
* Culture fails to meet specifications for study.
* Subject has any other medical condition that, in the opinion of the investigator, might significantly affect the ability to safely participate in the study or affect the conduct of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Is there any measurable effect upon the underlying cancer as assessed by an increase or decrease in the tumor as measured from baseline using established criteria? | 5 -15 Weeks

SECONDARY OUTCOMES:
Are the dosages administered during the study safe, as measured by the number of unexpected and serious adverse events associated with the study drug, as defined by FDA regulations and as measured by established criteria? | 5 - 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Korn, D.O., M.D., Principal Investigator — Envita Medical Centers
Locations (1):
- Envita Medical Centers, Scottsdale, Arizona, United States